CLINICAL TRIAL: NCT02396004
Title: Near-Infrared Red Spectroscopy (NIRS) to Measure Cerebral Perfusion During and After Patent Ductus Arteriosus (PDA) Treatment in Very Low Birth Weight (VLBW) Infants
Brief Title: NIRS in PDA VLBW Infants
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CIRB 2013/379/E
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: PDA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Near Infrared Red Spectroscopy (NIRS) — NIRS using INVOS cerebral/somatic oximeter

SUMMARY:
Aim of study:

To conduct an observational study to collect cerebral and renal perfusion data through NIRS before and after treatment of PDA by medication or by PDA ligation. The data post treatment would form the basis for normative baseline data in VLBW preterm newborn babies, particularly in the Asian population.

Study population/inclusion criteria:

VLBW newborn babies with hemodynamically significant PDA by echocardiography.

Exclusion criteria:

Major malformations Moribund patients

DETAILED DESCRIPTION:
Aim of study:

To conduct an observational study to collect cerebral and renal perfusion data through NIRS before and after treatment of PDA by medication or by PDA ligation. The data post treatment would form the basis for normative baseline data in VLBW preterm newborn babies, particularly in the Asian population.

Study population/inclusion criteria:

VLBW newborn babies with hemodynamically significant PDA by echocardiography.

Exclusion criteria:

Major malformations Moribund patients

Protocol:

Consent will be obtained from parents of eligible newborns before treatment of hemodynamic significant PDA. To attach cerebral and renal oximeter by NIRS to these VLBW infants with PDAs for until 24 hours post closure of PDA. Doppler ultrasound will be performed on anterior cerebral artery (ACA) and/or middle cerebral artery (MCA) artery and/or renal artery(RA) before PDA treatment and/or 24hours after PDA closure.This study aims to use one of the more popular neonatal/paediatrics NIRS machine, which is the INVOS cerebral/somatic oximeter

The same patient will hence form its own control after treatment. Echocardiographic follow-up or clinical assessment for closure of the PDA will be performed 24-48 hours after the course of medication or surgical closure.

ELIGIBILITY:
Inclusion Criteria:

* VLBW infants with hemodynamically significant PDA by echocardiography

Exclusion Criteria:

* Major malformation
* Moribund

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: VLBW (defined as birthweight less than 1500g) infants with hemodynamically significant PDA (patent ductus arteriosus) requiring treatment, either medical or surgical
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
cerebral oximetry | 2 years

SECONDARY OUTCOMES:
renal oximetry | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Woei Bing Poon, MRCPCH, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore